CLINICAL TRIAL: NCT06475612
Title: Using the Geriatric Trauma Outcome Score (GTOS) to Stratify the Mortality Risk of Adult Trauma Patients
Brief Title: Using the GTOS to Stratify the Mortality Risk of Adult Trauma Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202400775B0
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-05

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries | interventions — Death Domain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma Patients: The study cohort included 46,808 trauma patients from the Trauma Registry System, covering the period from 2009 to 2021. Of these, 40,068 were adult patients aged 20 years and older.
  Interventions: Other: Death; Other: Survival

INTERVENTIONS:
Other: Death — Mortality group.
Other: Survival — Survival group.

SUMMARY:
Trauma significantly impacts both short- and long-term health outcomes, resulting in substantial mortality. Early identification and risk stratification in trauma patients are crucial for timely medical interventions. The Geriatric Trauma Outcome Score (GTOS), designed by incorporating age, the Injury Severity Score (ISS), and the need for packed red blood cell transfusion, has emerged as a valuable prognostic tool for elderly trauma patients, but its applicability to general trauma patients remains underexplored.

ELIGIBILITY:
Inclusion Criteria:

* The study includes all patients aged equal to or over twenty who had trauma.

Exclusion Criteria:

* Patients with burns.
* Patients with hangings.
* Patients with drowning.
* Patients with with unavailable laboratory data.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort included 46,808 trauma patients from the Trauma Registry System, covering the period from 2009 to 2021 Of these, 41,131 were adult patients aged 20 years and older. After excluding patients with burns (n = 1,040), hanging injuries (n = 19), drowning (n = 3), and unavailable laboratory data (n = 1), a final study population of 40,068 patients was analyzed. Within this cohort, there were 818 deaths, and 39,250 patients survived.
Sampling Method: Non-Probability Sample
Enrollment: 40068 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Mortality outcome | Through hospital stay of patients, an average of 14 days.
  Mortality outcome of trauma patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan